CLINICAL TRIAL: NCT00342329
Title: Lupus Nephritis: Role of Environmental and Occupational Exposures
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999901154; 01-E-N154
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-03-07

CONDITIONS: Lupus Nephritis
Keywords: Case-Control; Hydrocarbons; Metals; Silica; Tobacco Smoke; Lupus Nephritis; Environmental Exposures; Occupational Exposures
MeSH Terms: conditions — Lupus Nephritis

SUMMARY:
The purpose of this study is to examine hormonal and environmental risk factors (and possible gene-environmental interactions) involved in the etiology of lupus nephritis. Our study will focus on exposures to occupational and environmental agents that have been linked to the development of systemic lupus erythematosus (SLE) or renal disease (e.g., silica dust, smoking). We will also assess potential gene environment interactions. We will examine these exposures in 100 patients with renal biopsy with documented proliferative or membraneous nephritis. We will compare exposures in the lupus nephritis patients to lupus patients who do not have nephritis and to normal controls who have participated in the Carolina Lupus Study. One hundred lupus nephritis patients (age 18 years or older, of both genders and all races) will be identified through the Glomerular Disease Collaborative Network (GDCN) Nephropathology database and participating nephrologists at the Medical University of South Carolina, Duke University Medical Center and the East Carolina Medical School.

DETAILED DESCRIPTION:
The purpose of this study is to examine hormonal and environmental risk factors (and possible gene-environmental interactions) involved in the etiology of lupus nephritis. Our study will focus on exposures to occupational and environmental agents that have been linked to the development of systemic lupus erythematosus (SLE) or renal disease (e.g., silica dust, smoking). We will also assess potential gene environment interactions. We will examine these exposures in 100 patients with renal biopsy with documented proliferative or membraneous nephritis. We will compare exposures in the lupus nephritis patients to lupus patients who do not have nephritis and to normal controls who have participated in the Carolina Lupus Study. One hundred lupus nephritis patients (age 18 years or older, of both genders and all races) will be identified through the Glomerular Disease Collaborative Network (GDCN) Nephropathology database and participating nephrologists at the Medical University of South Carolina, Duke University Medical Center and the East Carolina Medical School.

ELIGIBILITY:
* INCLUSION CRITERIA:

Have renal biopsy proven Lupus Nephritis (with the biopsy-based diagnosis date no earlier than January 1, 1995).

Reside within designated counties of eastern North Carolina and South Carolina.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0
Dates: Start 2001-04-16; Study Completion 2007-03-07

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of North Carolina, Chapel Hill, North Carolina
  - NIEHS, Research Triangle Park, Research Triangle Park, North Carolina